CLINICAL TRIAL: NCT03658603
Title: Thoracodorsal Artery Perforator Flap Versus Other Conventional Free Flaps in Soft Tissue Reconstruction
Brief Title: Thoracodorsal Artery Perforator Flap Versus Conventional Free Flaps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Diefy Salem, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAPF
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Thoracodorsal artery perforator flap
  Interventions: Procedure: thoracodorsal artery perforator flap
- control group (Active Comparator): Conventional free flaps
  Interventions: Procedure: latissimus dorsi flap

INTERVENTIONS:
Procedure: thoracodorsal artery perforator flap — fascio-cutaneous flap used in cases of trauma or burns
  Arms: Study group
Procedure: latissimus dorsi flap — musculo-cutaneous flap used in cases of trauma or burns
  Arms: control group

SUMMARY:
The purpose of this study is to assess the efficacy of the thoracodorsal artery perforator flap versus other conventional free flaps for reconstruction of soft tissue defects.

DETAILED DESCRIPTION:
The field of plastic surgery, unlike most other surgical specialties, has no anatomic or functional area to which it can lay claim; the plastic surgeon practices methods and techniques applicable to all specialties and anatomic areas.

Reconstructive surgery is the process of restoring the human body to "whole" following tumor extirpation, infection, trauma or congenital or acquired deformity - restoring both form and function.

The purpose of this study is to assess the efficacy of the thoracodorsal artery perforator flap versus other conventional free flaps for reconstruction of soft tissue defects.

ELIGIBILITY:
Inclusion Criteria:

• Soft tissue loss anywhere in the body.

Exclusion Criteria:

• Patients with chronic debilitating diseases e.g. chronic renal failure, uncontrolled diabetes mellitus

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-03 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
The mean operative time | 12 hours
  the time from the start to the end of operation

SECONDARY OUTCOMES:
The percentage of patients with Flap viability | 1 week
  The perforator flap will be assessed regarding (color, temperature, capillary refilling, congestion, blistering)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cannon B. The flowering of plastic surgery. JAMA. 1990 Feb 9;263(6):862-4. No abstract available. PMID 2404152
- [Background] Mardini S, Wei FC, Salgado CJ, Chen HC. Reconstruction of the reconstructive ladder. Plast Reconstr Surg. 2005 Jun;115(7):2174. doi: 10.1097/01.prs.0000165497.92397.be. No abstract available. PMID 15923904
- [Background] Lineaweaver WC. Microsurgery and the reconstructive ladder. Microsurgery. 2005;25(3):185-6. doi: 10.1002/micr.20125. No abstract available. PMID 15779080
- [Background] Geddes CR, Morris SF, Neligan PC. Perforator flaps: evolution, classification, and applications. Ann Plast Surg. 2003 Jan;50(1):90-9. doi: 10.1097/00000637-200301000-00016. PMID 12545116
- [Background] Wei FC, Mardini S. Free-style free flaps. Plast Reconstr Surg. 2004 Sep 15;114(4):910-6. doi: 10.1097/01.prs.0000133171.65075.81. PMID 15468398
- [Background] Hwang JH, Kim ES, Kim KS, Kim DY, Lee SY. Latissimus dorsi muscle and its short perforator-based skin compound free flap. Ann Plast Surg. 2007 Apr;58(4):381-7. doi: 10.1097/01.sap.0000243998.35882.7d. PMID 17413879
- [Background] Russell RC, Pribaz J, Zook EG, Leighton WD, Eriksson E, Smith CJ. Functional evaluation of latissimus dorsi donor site. Plast Reconstr Surg. 1986 Sep;78(3):336-44. doi: 10.1097/00006534-198609000-00009. PMID 3737758
- [Background] Wei FC, Jain V, Celik N, Chen HC, Chuang DC, Lin CH. Have we found an ideal soft-tissue flap? An experience with 672 anterolateral thigh flaps. Plast Reconstr Surg. 2002 Jun;109(7):2219-26; discussion 2227-30. doi: 10.1097/00006534-200206000-00007. PMID 12045540
- [Background] Kim JT, Koo BS, Kim SK. The thin latissimus dorsi perforator-based free flap for resurfacing. Plast Reconstr Surg. 2001 Feb;107(2):374-82. doi: 10.1097/00006534-200102000-00012. PMID 11214052
- [Background] Lin CT, Huang JS, Yang KC, Hsu KC, Chen JS, Chen LW. Reliability of anatomical landmarks for skin perforators of the thoracodorsal artery perforator flap. Plast Reconstr Surg. 2006 Nov;118(6):1376-1386. doi: 10.1097/01.prs.0000239525.44657.81. PMID 17051108
- [Background] Hallock GG. Direct and indirect perforator flaps: the history and the controversy. Plast Reconstr Surg. 2003 Feb;111(2):855-65; quiz 866. doi: 10.1097/01.PRS.0000040462.38363.C7. PMID 12560714